CLINICAL TRIAL: NCT04937413
Title: PEskE: A Phase 0/Surgical Window-of-opportunity Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Evolocumab in Patients With Recurrent High-grade Glioma or Glioblastoma
Brief Title: The PCSK9i Inhibitor Evolocumab - a Surgical Trial of Pharamcodynamics and Kinetics Evaluation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00108375
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Malignant Glioma; Glioblastoma
Keywords: Pro00108375; Khasraw; PCSK9i; Evolocumab; Glioma; Glioblastoma; PEskE
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single dose of evolocumab (Experimental): 420 mg of evolocumab subcutaneous injection 7-14 days before scheduled surgery for malignant glioma
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Evolocumab subcutaneous injection
  Other Names: Repatha

SUMMARY:
This Phase 0 surgical window of opportunity trial seeks to evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) properties of an FDA-approved proprotein convertase/ kexin type 9 serine protease inhibitor (PCSK9i) in patients with primary and recurrent World Health Organization (WHO) grade IV malignant glioma. The investigators intend to evaluate whether a clinically licensed PCSK9i called evolocumab (also known as Repatha) can be repurposed as a potential immunotherapeutic for high grade glioma by testing its ability to access the intracranial space. The primary objective is to evaluate whether evolocumab crosses the blood brain barrier (BBB) and is measurable in the resected tumor specimens of patients with primary and recurrent high grade glioma or glioblastoma.

DETAILED DESCRIPTION:
A maximum of 10 participants will receive 420 mg (the maximum single dose) of evolocumab subcutaneously into their thigh, abdomen or upper arm 7-14 days prior to surgical de-bulking of their tumor. After de-bulking, leftover tissue not required for histological analysis will be collected, and the level of evolocumab will be quantified. At two time points, prior to injection of evolocumab and at time of their surgery, participants will have peripheral blood drawn to analyze serum levels of the drug (for comparison to levels found in their leftover tissue). The investigators will follow-up with participants about 2 weeks after surgery at their post-operative visit.

A matched cohort of resected tumor specimens from patients who were not treated with evolocumab from the Duke Brain Tumor Center Biorepository will be used as a comparison for the primary objective and 2 of the 3 secondary objectives of this study comparing brain tumor tissue specimens of patients who did and did not receive evolocumab with respect to lipid metabolism and tumor cells expressing MHC-I.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Newly diagnosed or recurrent high grade glioma (HGG) or glioblastoma (GBM) (if recurrent, prior pathology report indicating HGG or GBM)
* Adequate hematologic function within 14 days prior to starting evolocumab defined as follows:

  1. Hemoglobin ≥ 10 g/dl (Note: the use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable)
  2. Leukocytes ≥ 1,500/mm3
  3. Absolute Neutrophil Count (ANC) ≥ 1,000/mm3
  4. Platelets ≥ 100,000/mm3
* Adequate renal function within 14 days prior to starting evolocumab defined as calculated creatinine clearance (CrCL) of ≥ 30 mL/min/1.73m2 by the Cockcroft-Gault formula
* Adequate hepatic function within 14 days prior to starting evolocumab defined as follows:

  1. Total bilirubin ≥ 1.5 x institutional upper limit of normal (ULN) (Note: Patients with known Gilbert disease without other clinically significant liver abnormalities are not excluded.)
  2. AST(SGOT) and ALT(SGPT) ≥ 1.5 × ULN
* Negative serum pregnancy test (in females of childbearing potential) within 48 hours of starting evolocumab.

Exclusion Criteria:

* Any patient with a history of a serious hypersensitivity reaction to evolocumab or any of the excipients in evolocumab
* Patients with severe hepatic impairment outside of the range defined in the inclusion criteria within 7 days of starting evolocumab.
* History or evidence of central nervous system bleeding as defined by stroke or intraocular bleed (including embolic stroke) not associated with any antitumor surgery within 6 months before enrollment
* Infection requiring intravenous antibiotics that was completed < 1 week of study enrollment (day 1) with the exemption of prophylactic antibiotics for long line insertion or biopsy
* Females of reproductive potential and males who are unwilling to practice an acceptable method(s) of effective birth control while on study through 1 month (2 half-lives) after receiving the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Presence of evolocumab in surgical tumor tissue and tissue from a matched control group | At time of surgical resection
  Determined by mass spectrometry

SECONDARY OUTCOMES:
Level of lipid metabolism within the surgical tumor tissue and tissue from a matched control group | At time of surgical resection
  Determined by fluorescence-activated cell sorting (FACS)
Major histocompatibility complex-1 (MHC-I) expression within the surgical tumor tissue and tissue from a matched control group | At time of surgical resection
  Determined by FACS
Correlation between serum and surgical tumor tissue levels of evolocumab | 2 weeks
  Using serum taken before receiving evolocumab (7-14 days before surgery) and serum taken at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04937413/Prot_SAP_000.pdf